CLINICAL TRIAL: NCT04605185
Title: Dose Escalation Study Of Donafenib and Toripalimab Combined With TACE in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Donafenib and Toripalimab Combined With TACE in Patients With Unresectable Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001D-C-103
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib/JS001/TACE (Experimental): Donafenib and JS001 Combined With TACE
  Interventions: Drug: Donafenib Tosilate Tablets; Biological: Toripalimab Injection

INTERVENTIONS:
Drug: Donafenib Tosilate Tablets — 100mg Qd/150mg Qd/100mg Bid, po
Biological: Toripalimab Injection — 240 mg, iv drip,q3w
  Other Names: JS001

SUMMARY:
This study is the single-center, open-label phase I clinical trial to evaluate tolerability, safety and efficacy of Donafenib and JS001 in combination with TCAE in patients with Unresectable Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
The phase I clinical trial is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of Donafenib in this regimen, and select an acceptable safe dose for the phase II clinical trial(RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 (inclusive), male or female;
* Diagnosis of Unresectable Hepatocellular Carcinoma confirmed clinically or histologically or cytologically according to the "Guidelines for diagnosis and treatment of primary liver cancer" (2019 Edition);
* At least one measurable lesion (according to RECIST v1.1)
* ECOG performance status score of 0 -1;
* Life expectancy ≥ 12 weeks;
* Fully understand this research and voluntarily sign the ICF.

Exclusion Criteria:

* Diffuse liver cancer；
* Refractory hepatic encephalopathy, refractory ascites, or hepatorenal syndrome；
* Pregnancy or lactation；
* Patients with extrahepatic diffusion；
* Spontaneous tumor rupture；
* Expected non-compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity(DLT) | 21 days after the first dose of JS001 and Donafenib, assessed up to 2 years
  Dose limiting toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity.

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization until death due to any cause, assessed up to 2 years.
  The Kaplan-Meier survival from the initiation date of first cycle until death from any cause or the last follow-up date.
Progression free survival (PFS) | From date of randomization until the date of objective disease progression or death, assessed up to 2 years.
  The Kaplan-Meier survival from the initiation date of first cycle until the date of first documented progression or date of death
Duration of response (DOR) | From the date of first documented response (RECIST 1.1.) until the first date of documented progression or death in the absence of disease progression, assessed up to 2 years.
  defined as the time between the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Shanzhi Gu, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No